CLINICAL TRIAL: NCT05224089
Title: Bilateral Mid-Abdominal Transverse Abdominis Plane and Rectus Sheath Blocks Comparing The Use of Liposomal Bupivacaine/Bupivacaine vs. Regular Bupivacaine in Laparoscopic Colectomy Procedures.
Brief Title: Bilateral TAP and RS Blocks Using Liposomal Bupivacaine/Bupivacaine vs. Regular Bupivacaine in Laparoscopic Colectomy
Acronym: TAPLIP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hartford Hospital (Other)
Responsible Party: Principal Investigator, Kevin Finkel, Director of Clinical Research - HH Department of Anesthesiology, Hartford Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HHC-2021-0331
Record Dates: First submitted 2021-11-17; First posted 2022-02-04 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Bowel Disease
Keywords: Liposomal Bupivacaine; Exparel; Bupivacaine; Laparoscopic Colectomy; Transverse Abdominis Plane Blocks (TAP); Regional anesthesia; Rectus Sheath Block
MeSH Terms: conditions — Intestinal Diseases | interventions — Bupivacaine; Dexamethasone; Epinephrine

STUDY DESIGN:
Intervention Model Description: single-center, prospective, triple blinded, randomized, controlled trial.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Triple (Participant, Care Provider, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Liposomal Bupivacaine/Bupivacaine HCL (Experimental): 20mL 1.3% Exparel (266mg) + 60mL 0.25% bupivacaine (150mg) + 20mL normal saline. Total 100mL divided into 10mL syringes, 30 mL left TAP, 30mL right TAP, 20mL left rectus, 20mL right rectus.
  Interventions: Drug: Liposomal Bupivicaine/Bupivacaine Admixture; Drug: Bupivacaine HCL
- Regular Bupivacaine Arm (Active Comparator): 80mL 0.25% bupivacaine (200mg) + 300mcg (0.3mL) epinephrine + 5mg (0.5mL) preservative free dexamethasone + 20mL of normal saline. Total 100mL divided into 10mL syringes, 30mL left TAP, 30mL right TAP, 20mL left rectus, 20mL right rectus.
  Interventions: Drug: Bupivacaine HCL

INTERVENTIONS:
Drug: Liposomal Bupivicaine/Bupivacaine Admixture — 60mL of 0.25% Bupivacaine (150mg)+ 20 mL of 1.3% Exparel (266 mg)+20mL NS=100mL
  Other Names: Bupivacaine
  Arms: Liposomal Bupivacaine/Bupivacaine HCL
Drug: Bupivacaine HCL — 80mL 0.25% bupivacaine (200mg) + 300mcg (0.3mL) epinephrine + 5mg (0.5mL) preservative free dexamethasone + 20mL NS= 100mL
  Other Names: Dexamethasone 0.5 ml (5 mg); Epinephrine 0.1 ml

SUMMARY:
This study will be a single center, prospective triple blinded randomized controlled study, comparing the use of liposomal bupivacaine (Exparel) to regular bupivacaine with adjuncts in bilateral mid-abdominal transverse abdominis plane (TAP) blocks for patients undergoing laparoscopic colectomy procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective laparoscopic colectomy surgery to be performed by one of the 4 colorectal surgeons in the study.
* English speaking patients
* Patients with American Society of Anesthesiology (ASA) physical status score I- IV

Exclusion Criteria:

1. Emergency laparoscopic colectomy surgery
2. Patients with distant metastatic cancers (e.g. bone, lung, brain).
3. Scheduled for multi organs resection surgery in addition to colectomy.
4. Patients with contraindications to TAP or RS blocks including but not limited to anatomical abnormality, previous surgical intervention that limits or prevents receiving bilateral TAP blocks (e.g. surgical mesh at the site of TAP or RS block), or infection at the injection site.
5. Current colostomies.
6. History of allergy to local anesthetics.
7. Coagulopathy or coagulation disorder. Also patients who are receiving antithrombotic medications as a contraindication to receiving single shot peripheral nerve blockade as per the most recent American Society of Regional Anesthesiology (ASRA) guidelines.16
8. Weight < 40 kg, as 40 mL of Bupivacaine 0.25%, or combination of 20 mL of bupivacaine 0.25% with 20 mL of liposomal bupivacaine is greater than the maximal dose allowed, given concern for local anesthetic toxicity.
9. Patients who take long acting opioid medication, or on continuous opioid > 50 MME per day for at least 30 days within 90 days prior to surgery. Also patients who have chronic pain syndrome with a recent preoperative consultation to the chronic pain service.
10. Patients with current substance abuse, or history of substance abuse within 3 months, this includes any illicit drugs or excessive alcohol consumption as defined 4 or more drinks per day or 8 or more drinks per week for women and 5 or more drinks per day or 15 or more drinks per week for men.15
11. Pregnant, nursing, or planning to become pregnant during the study or within 1 month postoperatively
12. Refusal or lack of providing the study consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2022-04-27 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
The highest Numerical Pain Scores | 3 days
  To compare the highest (worst) pain reported for the period of 48-72 hours post-surgery.

SECONDARY OUTCOMES:
The highest Numerical Pain Scores for the period of 0-47 hours | up to 3 days
  To compare the highest (worst) pain reported for the period of 48-72 hours post-surgery by patients in the two groups, using the Brief Pain Inventory (Short Form), this measurement will be done at the 26th and 50th postoperative hour with a range on +3/-2 hours.
All pain scores, mild-moderate-severe. | up to 72 postoperative hours
  Proportion of patients experiencing moderate or severe pain, the scores will be grouped such that 1-3 is considered mild pain, 4-6 moderate pain, and 7-10 severe pain.
Postoperative opioid consumption measured in morphine MilliEquivalent (MME) | Up to 6 days post surgery.
  Postoperative total opioid consumption measured in morphine MilliEquivalent (MME) will be collected starting from the time in post-anaesthesia care unit up to the first 6 postoperative days. Patients will continue to report their opioid consumption after discharge days using the pain and medication diary up to 6 days post-surgery.
Postoperative nausea/vomiting scores | 30 days
  Using a validated measure; the Simplified (Post-operative nausea and vomiting Impact Scale 17 which consists of two questions, each with a possible response score of 0-3. Response score totals of 0-2 require no intervention. Response score totals of 3-4 may necessitate antiemetic medication. Response score totals of 5-6 are considered clinically important nausea requiring medication intervention, as this would constitute patients with excessive vomiting. This form will be completed either by the assigned nurse or the study coordinator immediately after surgery in the post-anesthesia care unit, postoperative day#1, postoperative day#2, postoperative day#3, and during the first follow up visit.
Hospital and post-anesthesia care unit length of stay | 6 days
  Hospital length of stay will be calculated in hours from the date and time of admission and discharge from the electronic medical records. post-anesthesia care unit length of stay will be calculated in minutes using the post-anesthesia care unit data collection sheet and from the electronic medical records.
Duration of the study block using the sensory function test | Pre-block intervention, immediately after surgery, up to 3 days
  The preoperative sensory function test will be assessed prior to the block by the anesthesiologist performing the block while the postoperative assessment at the post-anesthesia care unit will be used as baseline to be compared with the following sensory tests to assess the duration of sensory nerve block, using post-anesthesia care unit and In-Patient Post-Operative Data Collection Sheet.
Brief Pain Inventory (Short Form) | On the day of first postoperative visit, the end of the 6th and 12th postoperative months
  A validated scale that rapidly assesses pain severity and its impact on functioning. It consists of a 2-page questionnaire that asks patients to report the location and severity of their pain, and to report the interference of pain, if any, on their activities over the previous 24 hours. Four questions ask patients to rate the severity of their pain on a scale of 1-10 over the previous 24 hours in 4 discrete categories: worst, least, average, and right now. Each rating is analyzed separately. Seven questions ask patients to rate how severely their pain has interfered with their general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life on a scale of 1-10 over the previous 24 hours. These 7 questions are scored as a mean of the answers given, as long as at least 4 questions are answered. Two other questions ask patients to list the treatments or medications they are currently using, and to rate how much relief these are providing.
Block complications | Up to 30 postoperative days
  The occurrence of block complications will be collected intraoperative and postoperative period including post-anesthesia care unit, daily in patient period, the day of discharge, and at the time of the post-operative follow-up visit. Readmissions within 30 days after discharge will also be collected.
Patient Overall Satisfaction | 30 days
  A scale from 0 = very dissatisfied to 10 = very satisfied, this will be evaluated on day of discharge and on the first postoperative clinic visit either in person or through a phone call.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Finkel, MD, Principal Investigator — Hartford Hospital
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim AJ, Yong RJ, Urman RD. The Role of Transversus Abdominis Plane Blocks in Enhanced Recovery After Surgery Pathways for Open and Laparoscopic Colorectal Surgery. J Laparoendosc Adv Surg Tech A. 2017 Sep;27(9):909-914. doi: 10.1089/lap.2017.0337. Epub 2017 Jul 25. PMID 28742435
- [Background] Varadhan KK, Neal KR, Dejong CH, Fearon KC, Ljungqvist O, Lobo DN. The enhanced recovery after surgery (ERAS) pathway for patients undergoing major elective open colorectal surgery: a meta-analysis of randomized controlled trials. Clin Nutr. 2010 Aug;29(4):434-40. doi: 10.1016/j.clnu.2010.01.004. Epub 2010 Jan 29. PMID 20116145
- [Background] Stokes AL, Adhikary SD, Quintili A, Puleo FJ, Choi CS, Hollenbeak CS, Messaris E. Liposomal Bupivacaine Use in Transversus Abdominis Plane Blocks Reduces Pain and Postoperative Intravenous Opioid Requirement After Colorectal Surgery. Dis Colon Rectum. 2017 Feb;60(2):170-177. doi: 10.1097/DCR.0000000000000747. PMID 28059913
- [Background] Fields AC, Weiner SG, Maldonado LJ, Cavallaro PM, Melnitchouk N, Goldberg J, Stopfkuchen-Evans MF, Baker O, Bordeianou LG, Bleday R. Implementation of liposomal bupivacaine transversus abdominis plane blocks into the colorectal enhanced recovery after surgery protocol: a natural experiment. Int J Colorectal Dis. 2020 Jan;35(1):133-138. doi: 10.1007/s00384-019-03457-1. Epub 2019 Dec 4. PMID 31797098
- [Background] Smith SR, Draganic B, Pockney P, Holz P, Holmes R, Mcmanus B, Carroll R. Transversus abdominis plane blockade in laparoscopic colorectal surgery: a double-blind randomized clinical trial. Int J Colorectal Dis. 2015 Sep;30(9):1237-45. doi: 10.1007/s00384-015-2286-7. Epub 2015 Jun 24. PMID 26099316
- [Background] Qazi N, Bhat WM, Iqbal MZ, Wani AR, Gurcoo SA, Rasool S. Postoperative Analgesic Efficacy of Bilateral Transversus Abdominis Plane Block in Patients Undergoing Midline Colorectal Surgeries Using Ropivacaine: A Randomized, Double-blind, Placebo-controlled Trial. Anesth Essays Res. 2017 Jul-Sep;11(3):767-772. doi: 10.4103/0259-1162.194577. PMID 28928585
- [Background] Erratum to highlighted version successful resection of a tracheal metastasis of rectal cancer: a case report. J Thorac Dis. 2017 Oct;9(10):E978. doi: 10.21037/jtd.2017.10.137. PMID 29266106
- [Background] Liu L, Xie YH, Zhang W, Chai XQ. Effect of Transversus Abdominis Plane Block on Postoperative Pain after Colorectal Surgery: A Meta-Analysis of Randomized Controlled Trials. Med Princ Pract. 2018;27(2):158-165. doi: 10.1159/000487323. Epub 2018 Feb 1. PMID 29402875
- [Background] Chahar P, Cummings KC 3rd. Liposomal bupivacaine: a review of a new bupivacaine formulation. J Pain Res. 2012;5:257-64. doi: 10.2147/JPR.S27894. Epub 2012 Aug 14. PMID 23049275
- [Background] Keller DS, Tahilramani RN, Flores-Gonzalez JR, Ibarra S, Haas EM. Pilot study of a novel pain management strategy: evaluating the impact on patient outcomes. Surg Endosc. 2016 Jun;30(6):2192-8. doi: 10.1007/s00464-015-4459-4. Epub 2015 Aug 15. PMID 26275549
- [Background] Hutchins JL, Kesha R, Blanco F, Dunn T, Hochhalter R. Ultrasound-guided subcostal transversus abdominis plane blocks with liposomal bupivacaine vs. non-liposomal bupivacaine for postoperative pain control after laparoscopic hand-assisted donor nephrectomy: a prospective randomised observer-blinded study. Anaesthesia. 2016 Aug;71(8):930-7. doi: 10.1111/anae.13502. Epub 2016 May 30. PMID 27238859
- [Background] Hutchins J, Argenta P, Berg A, Habeck J, Kaizer A, Geller MA. Ultrasound-guided subcostal transversus abdominis plane block with liposomal bupivacaine compared to bupivacaine infiltration for patients undergoing robotic-assisted and laparoscopic hysterectomy: a prospective randomized study. J Pain Res. 2019 Jul 4;12:2087-2094. doi: 10.2147/JPR.S193872. eCollection 2019. PMID 31308734
- [Background] Hozo SP, Djulbegovic B, Hozo I. Estimating the mean and variance from the median, range, and the size of a sample. BMC Med Res Methodol. 2005 Apr 20;5:13. doi: 10.1186/1471-2288-5-13. PMID 15840177
- [Background] Wan X, Wang W, Liu J, Tong T. Estimating the sample mean and standard deviation from the sample size, median, range and/or interquartile range. BMC Med Res Methodol. 2014 Dec 19;14:135. doi: 10.1186/1471-2288-14-135. PMID 25524443
- [Background] Horlocker TT, Vandermeuelen E, Kopp SL, Gogarten W, Leffert LR, Benzon HT. Regional Anesthesia in the Patient Receiving Antithrombotic or Thrombolytic Therapy: American Society of Regional Anesthesia and Pain Medicine Evidence-Based Guidelines (Fourth Edition). Reg Anesth Pain Med. 2018 Apr;43(3):263-309. doi: 10.1097/AAP.0000000000000763. No abstract available. PMID 29561531
- [Background] Myles PS, Wengritzky R. Simplified postoperative nausea and vomiting impact scale for audit and post-discharge review. Br J Anaesth. 2012 Mar;108(3):423-9. doi: 10.1093/bja/aer505. Epub 2012 Jan 29. PMID 22290456
- [Background] Liang M, Xv X, Ren C, Yao Y, Gao X. Effect of ultrasound-guided transversus abdominis plane block with rectus sheath block on patients undergoing laparoscopy-assisted radical resection of rectal cancer: a randomized, double-blind, placebo-controlled trial. BMC Anesthesiol. 2021 Mar 24;21(1):89. doi: 10.1186/s12871-021-01295-9. PMID 33761901
- [Background] Nagata J, Watanabe J, Sawatsubashi Y, Akiyama M, Arase K, Minagawa N, Torigoe T, Hamada K, Nakayama Y, Hirata K. A novel transperitoneal abdominal wall nerve block for postoperative pain in laparoscopic colorectal surgery. Asian J Surg. 2018 Sep;41(5):417-421. doi: 10.1016/j.asjsur.2017.02.006. Epub 2017 Apr 25. PMID 28389063
- [Background] Tor, I.H., Çelik, E.C. & Aydın, M.E. Analgesic effect of combined transversus abdominis plane block and rectus sheath block in laparoscopic cholecystectomy: prospective randomized study. Ain-Shams J Anesthesiol 12, 58 (2020). https://doi.org/10.1186/s42077-020-00108-4
- [Background] Connolly NC. Real-world insights on the use of transversus abdominis plane block with liposomal bupivacaine in the multimodal management of somatic versus visceral pain in the colorectal surgery setting. J Pain Res. 2018 Jun 15;11:1141-1146. doi: 10.2147/JPR.S168817. eCollection 2018. No abstract available. PMID 29942149